CLINICAL TRIAL: NCT00271323
Title: A Two Arm Phase II Study Assessing Docetaxel/Cisplatin Induction Therapy Followed by Concurrent Chemoradiotherapy or Concurrent Chemoradiotherapy Followed by Consolidation Docetaxel/Cisplatin in Patients With Locally Advanced Unresectable NSCLC (Stage IIIA-multiple cN2 or IIIB)
Brief Title: Safety Study of Docetaxel/Cisplatin Induction Therapy Followed by Concurrent Chemoradiotherapy or Concurrent Chemoradiotherapy Followed by Consolidation Docetaxel/Cisplatin in NSCLC Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: "Medical Affairs Study Director", sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976B_2507; EudraCT #: 2005-001276-12
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Induction chemotherapy followed by concurrent chemoradiotherapy
  Interventions: Drug: docetaxel and cisplatin
- 2 (Active Comparator): Concurrent chemo-radiotherapy followed by consolidation chemotherapy
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: docetaxel and cisplatin — Docetaxel (75 mg/m2, IV, Day 1) and cisplatin (40 mg/m2, IV, Day 1, 2) every 3 weeks for 2 cycles, followed by concurrent chemo-radiotherapy with docetaxel (20 mg/m2, IV) and cisplatin (20 mg/m2) weekly for 6 weeks + radiotherapy 2 Gy/day, 5 days per week to a total dose of 66 Gy.
  Arms: 1
Radiation: radiotherapy — Docetaxel (20 mg/m2, IV) and cisplatin (20 mg/m2) weekly for 6 weeks + radiotherapy 2 Gy/day, 5 days per week to a total dose of 66 Gy followed by docetaxel (75 mg/m2, IV, Day 1) and cisplatin (40 mg/m2, IV, Day 1, 2) every 3 weeks for 2 cycles.
  Arms: 2

SUMMARY:
* Primary : To determine the safety profile of each treatment group.
* Secondary : To determine efficacy in term of overall response, disease free survival and survival at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form obtained, signed and dated before specific protocol procedures.
2. Histologically or cytologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma or a combination of these)
3. Patients must have a loco regionally advanced unresectable NSCLC;

   * Stage IIIA with clinical multiple N2 nodes (preferably with histological or cytological confirmation).

     * Patients with peripheral tumours of the lower lobe with contralateral upper mediastinal nodes at station N2 are excluded·
   * Stage IIIB T4 or N3.

     * In the T4 category, patients with pleural or pericardial effusion and multiple nodules in the same lobe are excluded.
     * Patients with T4 disease secondary to extensive and massive involvement of the great vessels are excluded.Patients should be excluded when the expected risk of pulmonary toxicity is likely to be high, e.g. V20 in excess of 35%.
4. Males or females aged between 18 and 75 years.
5. Life expectancy of at least 12 weeks.
6. WHO performance status 0 or 1.
7. Weight loss <=10% within the last 3 months.
8. Laboratory requirements at entry (within 7 days before randomization):

   * Blood cell counts:

     * Absolute neutrophils >= 2.0 x 10^9/L
     * Platelets >= 100 x 10^9/L
     * Hemoglobin >= 10 g/dl
   * Renal function:

     * Serum creatinine <=1 x the upper limit of normal (UNL). In case of borderline value of serum creatinine, the 24h creatinine clearance should be >= 60 mL/min.
   * Hepatic function:

     * Serum bilirubin <= 1 x UNL
     * ASAT and ALAT <= 2.5 x UNL
     * Alkaline phosphatase <= 5 x UNL Patients with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase> 2.5 x UNL are not eligible for the study.
9. Lung function tests at entry:

   * FEV1: >= 50 % x Normal value
   * DLCO: >= 50 % x Normal value
10. Adequate cardiac function.
11. Patient with either measurable and/or non-measurable lesion (according to RECIST criteria).

Exclusion Criteria:

1. Diagnosis of small cell lung cancer.
2. Pregnant or lactating women.
3. Patients (male or female) with reproductive potential not implementing adequate contraceptive measures.
4. Prior systemic chemotherapy, immunotherapy, or biological therapy including neoadjuvant or adjuvant treatment for NSCLC.
5. Prior surgery for NSCLC, if less than 5 years from study.
6. Prior radiotherapy for NSCLC.
7. History of prior malignancies, except for cured non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years.
8. Symptomatic peripheral neuropathy Grade >= 2 except if due to trauma.
9. Other serious concomitant illness or medical conditions:

   * Congestive heart failure or angina pectoris except if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmias.
   * History of significant neurological or psychiatric disorders including dementia or seizures.
   * Active infection requiring IV antibiotics.
   * Active ulcer, unstable diabetes mellitus or other contra-indication to corticosteroid therapy.
   * Superior vena cava syndrome contra-indicating hydration.
   * Preexisting pericardial effusion.
   * Preexisting symptomatic pleural effusion.
10. Significant gastrointestinal abnormalities, including requirement for intravenous nutrition, active peptic ulcer disease, prior surgical procedures affecting absorption.
11. Distant metastasis.
12. Concurrent treatment with any other experimental anti-cancer drugs.
13. Concomitant or within 4-week period administration of any other experimental drug under investigation.
14. Significant ophthalmologic abnormalities.
15. Moderate to severe dermatitis.
16. Hypersensitivity to docetaxel, cisplatin, or any of its excipients.
17. Concomitant use of phenytoin, carbamazepin, barbiturates, or rifampicin.
18. Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
19. Patient unlikely to comply with protocol, i.e., uncooperative attitude, inability to return for follow-up visits, and not likely to complete the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
overall response rate | in population of patients eligible and evaluable for response
time to progression | from the date of start treatment until progression
duration of response | only on responders

CONTACTS AND LOCATIONS:
Overall Officials: M COUDERC, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France